CLINICAL TRIAL: NCT00416572
Title: Adjustment to Breast Cancer Among Younger Women
Brief Title: Educational Program in Younger Women Who Have Recently Finished Treatment for Stage I or Stage II Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michael F. Scheier, Professor of Psychology, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMU-00000603; 5R01CA064711 (NIH)
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Results first posted 2016-11-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-09

CONDITIONS: Breast Neoplasms
Keywords: psychosocial effects of cancer and its treatment; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Education Intervention (Experimental): Participants attended 4 2-hr education sessions. The overall goal of the sessions was to provide information that would reduce participants' uncertainty about their illness and its treatment, to enhance coping in productive ways with the issues and problems confronting them, and to facilitate communication between the participants and their partners.
  Interventions: Behavioral: Education Intervention
- Nutrition Education Intervention (Experimental): Participants attended 4 2-hr nutrition education sessions. Each session provided information and encouragement on setting and attaining measurable goals for healthy eating and on the benefits of thinking positively about dealing adaptively with problems in life and living a healthy lifestyle.
  Interventions: Behavioral: Nutrition Education Intervention
- Control Condition (No Intervention): Participants received care as usual.

INTERVENTIONS:
Behavioral: Education Intervention — Sessions were led by two professionals with expertise in the topic. The sessions began a with presentation of informational material followed by guided discussion of related topics. The first session discussed what to say and not say to children about cancer and how to create a safe environment for them; the second session discussed carrying on with life after the diagnosis of breast cancer, including strategies for managing stress and anxiety and developing meaning in life; the third session talked about how to maintain closeness with a partner and ways to talk about breast cancer; the last session focused on the effects of treatment on reproductive status, and the genetic bases of breast cancer. Participants were also given related booklets and brochures to take home to read.
  Arms: Education Intervention
Behavioral: Nutrition Education Intervention — The nutrition sessions were presented by a professional trained in nutritional science. Sessions included the presentation of information and guided discussion of related topics. The first session discussed information on choosing fruits, vegetables, and low-fat foods and incorporating them into a diet; the second session involved a demonstration of low-fat cooking methods; the third session provided information on the nutritional make-up of a healthy diet and how to shop for it; the last session included information on how to maintain a healthy, low-fat diet while eating out. Women were also asked to keep a four-day food diary, to focus them on their dietary intake and control over it.
  Arms: Nutrition Education Intervention

SUMMARY:
RATIONALE: Educational programs may improve coping and quality of life in younger women who have recently been treated for early-stage breast cancer.

PURPOSE: To conduct a clinical trial to determine if an educational intervention and a nutritional intervention could enhance physical and psychological functioning among younger women completing treatment for early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Design, implement, and evaluate an educational intervention and a nutrition education intervention specifically aimed at improving adjustment among younger women who have been newly diagnosed with and treated for stage I or II breast cancer and who are ending the active phase of treatment.
* Determine the processes through which the interventions affect quality of life.
* Assess whether the interventions are differentially effective for different groups of women.
* Determine how women who decline participation differ from those who participate.
* Determine the nature and extent of adjustment difficulties, using baseline data, in younger women living in an urban setting who have been treated for early stage breast cancer.
* Identify personality and situational correlates of individuals who adapt well to early-stage breast cancer diagnosis and treatment and those who do not.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 intervention groups or a control condition.

* Arm I (control group): Patients did not undergo any intervention. Patients were evaluated at baseline and at 4 and 13 months.
* Arm II (breast cancer education group): Patients attended a series of approximately 2-hour-long breast cancer education group sessions once a month for 4 months. Sessions involved the presentation of information concerning breast cancer, followed by a guided discussion of related topics. Sessions topics included: talking with children about cancer, life after diagnosis, relationships/intimacy, and hormones and breast cancer/basic factors of heredity. Patients were also given booklets and brochures to read at home. Patients were evaluated at baseline, immediately after the intervention, and at 9 months after the intervention.
* Arm III (nutritional education group): Patients attended a series of approximately 2-hour-long nutritional education group sessions once a month for 4 months. Sessions involved the presentation of information concerning nutrition, followed by a guided discussion of related topics. Session topics included: healthy cupboards, what's cooking, shopping for success, and out on the town. Patients were also asked to keep a 4 day record of diet. Patients were evaluated at baseline, immediately after the intervention, and at 9 months after the intervention.

ELIGIBILITY:
INCLUSION CRITERIA (Disease Characteristics):

* Diagnosis of breast cancer

  * Stage I or II disease
  * No more than 10 positive lymph nodes
  * First-time diagnosis
  * Under the age of 50 at diagnosis
* Finished active treatment within the past 2 months
* English-speaking only
* Must live within 30 miles of Magee Women's Hospital, Pittsburgh, Pennsylvania

INCLUSION CRITERIA (Patient Characteristics):

* Female patients only
* Must be able to communicate

EXCLUSION CRITERIA (Patient Characteristics):

* Other prior malignancies except skin cancer

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Actual)
Dates: Start 1997-01; Primary Completion 2001-05 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Scheier, PhD, Study Chair — Pittsburgh Mind-Body Center at Carnegie Mellon University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants were identified through nurse referrals of consecutive and potentially eligible patients from hospital medical oncology clinics and physicians' offices in southwestern Pennsylvania.
Groups:
- Education Intervention: Participants attended 2-hr education sessions once a month, for 4 months. The overall goal of the sessions was to provide information that would reduce participants' uncertainty about their illness/treatment, to enhance coping in productive ways.
  Sessions were led by two professionals with expertise in the topic. The sessions began a with presentation of informational material followed by guided discussion of related topics. The first session discussed what to say and not say to children about cancer; the second session discussed carrying on with life after the diagnosis of breast cancer, including strategies for managing stress and anxiety and developing meaning in life; the third session talked about how to maintain closeness with a partner and ways to talk about breast cancer; the last session focused on the effects of treatment on reproductive status, and the genetic bases of breast cancer. Participants were also given related booklets and brochures to take home to read.
- Nutrition Education Intervention: Participants attended 2-hr nutrition education sessions, once a month for 4 months. Each session provided information/ encouragement on setting and attaining goals for healthy eating and on the benefits of thinking positively about dealing adaptively with problems and living a healthy lifestyle.
  The nutrition sessions were presented by a professional trained in nutritional science. Sessions included the presentation of information and guided discussion of related topics. The first session discussed information on choosing fruits, vegetables, and low-fat foods and incorporating them into a diet; the second session involved a demonstration of low-fat cooking methods; the third session provided information on the nutritional make-up of a healthy diet and how to shop for it; the last session included information on how to maintain a healthy, low-fat diet while eating out. Women were also asked to keep a four-day food diary, to focus them on their dietary intake and control over it.
Period: Overall Study
Arm/Group | Education Intervention | Nutrition Education Intervention | Control Condition
Started | 83 | 85 | 84
Completed | 70 | 78 | 76
Not Completed | 13 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Education Intervention: Participants attended 2-hr education sessions once a month, for 4 months. The overall goal of the sessions was to provide information that would reduce participants' uncertainty about their illness/treatment, to enhance coping in productive ways.
- Nutrition Education Intervention: Participants attended 2-hr nutrition education sessions, once a month for 4 months. Each session provided information/ encouragement on setting and attaining goals for healthy eating and on the benefits of thinking positively about dealing adaptively with problems and living a healthy lifestyle.
- Total: Total of all reporting groups
Arm/Group | Education Intervention | Nutrition Education Intervention | Control Condition | Total
Number analyzed (Participants) | 83 | 85 | 84 | 252
Age, Continuous [Mean (Full Range); unit: years] | 43.7 [18 to 50] | 44.2 [18 to 50] | 44.6 [18 to 50] | 44.2 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 85 | 84 | 252
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 79 | 80 | 82 | 241
  African-American | 4 | 3 | 2 | 9
  Other | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms (Measured With an Abbreviated 10-item CES-D) at Baseline, Post-intervention (4-months Post-intervention) and Final Follow-up (13-months Post-intervention).
Description: Scores for the shortened form of the Center for Epidemiologic Studies Depression scale(CES-D) ranged from 0 (no depressive symptoms) to 24 (high levels of depressives symptoms) in the present sample.
Time Frame: Baseline, Post-intervention(4 months post-intervention) and Final Follow-up(13 months post-intervention).
Population: All women who agreed to random assignment and completed all three assessments were retained in the analysis regardless of their level of group attendance.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Intervention | Nutrition Education Intervention | Control Condition
Number analyzed (Participants) | 70 | 78 | 76
units on a scale
  Baseline | 5.83 (5.32) | 6.74 (5.94) | 6.70 (5.84)
  Post-intervention | 5.65 (5.53) | 5.70 (5.45) | 6.87 (5.84)
  Final follow-up | 5.07 (4.99) | 4.36 (4.49) | 6.88 (6.19)
Statistical Analysis 1: Comparison: Education Intervention vs Control Condition; Comparison between education intervention and the control condition at 4 months post-intervention. The full regression model contained 2 dummy-coded variables (education intervention vs. control condition and nutrition education intervention vs. control condition), and the baseline measure of the outcome; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 2: Comparison: Nutrition Education Intervention vs Control Condition; Comparison between nutrition education intervention and the control condition at 4 months post-intervention. The full regression model contained 2 dummy-coded variables (education intervention vs. control condition and nutrition education intervention vs. control condition), and the baseline measure of the outcome; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 3: Comparison: Education Intervention vs Control Condition; Comparison between education intervention and the control condition at final follow-up (13 months post-intervention). The full regression model contained 2 dummy-coded variables (education intervention vs. control condition and nutrition education intervention vs. control condition), and the baseline measure of the outcome; Test type: Superiority or Other; p = 0.08, Regression, Linear; standardized beta = -0.12
Statistical Analysis 4: Comparison: Nutrition Education Intervention vs Control Condition; Comparison between nutrition education intervention and the control condition at final follow-up (13 months post-intervention). The full regression model contained 2 dummy-coded variables (education intervention vs. control condition and nutrition education intervention vs. control condition), and the baseline measure of the outcome; Test type: Superiority or Other; p < 0.001, Regression, Linear; standardized beta = -0.23

2. Primary Outcome: Perceived Physical Health (Measured With SF-36) at Baseline, Post-intervention (4-months Post-intervention) and Final Follow-up (13-months Post-intervention)
Description: The Perceived Physical Health Component scale of the Medical Outcomes Study Short Form 36 (SF-36) consists of a norm-based weighted average of the following subscales: Physical functioning, bodily pain, role limitations due to physical problems and general health. In the present study, scores ranged from a maximum of 68 (high levels of perceived health) to a minimum of 24 (low levels of perceived health).
Time Frame: Baseline, Post-intervention(4 months post-intervention), and Final Follow-up(13 months post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Intervention | Nutrition Education Intervention | Control Condition
Number analyzed (Participants) | 70 | 78 | 76
units on a scale
  Baseline | 49.21 (8.19) | 50.38 (8.26) | 49.16 (8.26)
  Post-intervention | 52.03 (7.02) | 53.59 (6.18) | 50.73 (9.07)
  Final follow-up | 55.11 (7.12) | 53.90 (5.55) | 50.93 (9.14)
Statistical Analysis 1: Comparison: Education Intervention vs Control Condition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > 0.50, Regression, Linear
Statistical Analysis 2: Comparison: Nutrition Education Intervention vs Control Condition; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.04, Regression, Linear; Standardized beta = 0.14
Statistical Analysis 3: Comparison: Education Intervention vs Control Condition; Comparison between the education intervention and the control condition at final follow-up (13 months post-intervention). The full regression model contained 2 dummy-coded variables (education intervention vs. control condition and nutrition education intervention vs. control condition), and the baseline measure of the outcome; Test type: Superiority or Other; p < 0.001, Regression, Linear; Standardized beta = 0.25
Statistical Analysis 4: Comparison: Nutrition Education Intervention vs Control Condition; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p = 0.02, Regression, Linear; Standardized beta = 0.15

3. Primary Outcome: Mental Health (Measured With the SF-36) at Baseline, Post-intervention (4-months Post-intervention) and Final Follow-up (13-months Post-intervention)
Description: The Mental Health Component Scale of the Medical Outcomes Study Short Form 36 (SF-36) consists of a norm-based weighted average of the following subscales: vitality, social functioning, role limitations due to emotional problems and mental health. In the present study, scores ranged from a maximum of 68 (high levels of mental health) to a minimum of 15 (low levels of mental health).
Time Frame: Baseline, Post-intervention(4 months post-intervention), Final Follow-up(13 months post-intervention)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Education Intervention | Nutrition Education Intervention | Control Condition
Number analyzed (Participants) | 70 | 78 | 76
units on a scale
  Baseline | 45.63 (10.77) | 46.91 (11.18) | 45.76 (10.69)
  Post-Intervention | 50.47 (9.13) | 50.38 (9.06) | 49.27 (9.06)
  Final Follow-up | 48.64 (10.72) | 51.26 (8.27) | 49.48 (8.27)
Statistical Analysis 1: Comparison: Education Intervention vs Control Condition; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p > .05, Regression, Linear
Statistical Analysis 2: Comparison: Nutrition Education Intervention vs Control Condition; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 3: Comparison: Education Intervention vs Control Condition; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p > 0.05, Regression, Linear
Statistical Analysis 4: Comparison: Nutrition Education Intervention vs Control Condition; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p > 0.05, Regression, Linear

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Education Intervention | Nutrition Education Intervention | Control Condition
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/85 | 0/84
Other Adverse Events (participants affected / at risk) | 0/83 | 0/85 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No